CLINICAL TRIAL: NCT06416124
Title: Anthropometric Characteristics of Elite and Olympic Mexican Track and Field Athletes
Acronym: ANTHROLYMPMX
Status: Completed | Type: Observational
Sponsor: Iberoamerican Institute of Sports Science and Human Movement (Other)
Collaborators: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Cesar Octavio Ramos Garcia, PhD, Principal Investigator, Iberoamerican Institute of Sports Science and Human Movement
Other Study IDs: IICDEM-ID-001-2013
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Athletes
Keywords: Athletes; Kinanthropometry; Body composition; Somatotype; High performance; Track and Field

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite and Olympic Mexican track and field athletes: All 74 athletes competing in track and field events during the XXIV Central American and Caribbean Athletics Championship will be considered
  Interventions: Diagnostic Test: Anthropometric assessment

INTERVENTIONS:
Diagnostic Test: Anthropometric assessment — A total of 43 anthropometric variables (complete profile) will be assessed following the guidelines of the International Society for the Advancement of Kinanthropometry. All measurements will be taken on the right side of the body. The full anthropometric profile will be undertaken in duplicate to establish retest reliability. If the difference between duplicate measures exceeds 5% for skinfolds or 1% for all other variables, a third measurement will be taken, but only after the full profile has been completed in duplicate. The mean of duplicate or median of triplicate anthropometric measurements will be used for all subsequent analysis. The intra-evaluator technical error of measurement (TEM) was calculated according to the 1996 protocol of Pederson and Gore.

SUMMARY:
Sport specialization requires an understanding of morphological variability to optimize performance. However, the current literature lacks a detailed analysis of the anthropometric profile of track and field athletes, especially in Latin America. Additionally, the five-way fractionation method of body mass has been under-documented. These gaps highlight the need for more research to maximize the potential of athletes, particularly in emerging countries like Mexico. This study aims to determine the anthropometric characteristics of elite and Olympic Mexican track and field athletes. A descriptive cross-sectional study will be conducted. Forty-three anthropometric variables will be assessed to characterize the athlete´s physical composition using the standards of the International Society for the Advancement of Kinanthropometry (ISAK). Those variables will be used to describe the anthropometric profile (Heath and Carter somatotype, body composition through five-way fractionation method, muscle bone index, muscular adipose index, sum of skinfold thicknesses, and proportionality through Ross & Wilson Phantom strategy. Correspondences of those variables will also be established among different tests and specialties: sprint, middle-distance, long-distance, endurance, combined events, jumps, and throws. This study aims to provide the opportunity to generate reliable references for high-performance Mexican athletes.

ELIGIBILITY:
Inclusion Criteria:

* Elite and Olympic Mexican track and field athletes
* Female and male,
* All national teams
* Actively competing in national and/or international competitions

Exclusion Criteria:

* Injured or not classified athletes
* Not informed consent signed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Elite and Olympic Mexican track and field athletes from different national teams and actively competing in national and international competitions
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-07-05 (Actual); Primary Completion 2013-07-07 (Actual); Study Completion 2013-07-07 (Actual)

PRIMARY OUTCOMES:
Anthropometric body composition profile | One day
  Body composition assessment through anthropometric five-way fractionation method of Ross and Kerr

SECONDARY OUTCOMES:
Heath and Carter somatotype | One day
  A cuantitative method to assess body shape obtained from diferent anthropometric measurements
Anthropometric profile | One day
  A total of 43 measurements will be obtained using the standards of the methodology of the International Society for the Advancement of Kinanthropometry (ISAK)
Muscle Bone Ratio | One day
  Ratio between muscle mass and bone mass in Kg
Muscular Adipose Ratio | One day
  Ratio between muscle mass and adipose mass in Kg
Sum of skinfold thicknesses | One day
  Sum of 6 different skinfold thicknesses
Corrected girths | One day
  Correction of girth value by sustracting the skinfold thickness value
Proportionality | One day
  Ross phantom strategy for the analisys of body proportions

CONTACTS AND LOCATIONS:
Overall Officials: Wiliam Carvajal-Veitía, PhD, Principal Investigator — Institute of Sports Medicine (IMD), Cuba; Fernando Alacid-Carceles, PhD, Principal Investigator — University of Almeria (UAL), Spain; Rodrigo Yáñez-Sepúlveda, PhD, Principal Investigator — Andres Bello University (UNAB), Chile
Locations (1):
- Iberoamerican Institute of Sports Science and Human Movement, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Because the participants were informed that data management would be protected only by the principal investigators.

REFERENCES:
- [Background] Bernal-Orozco MF, Posada-Falomir M, Quinonez-Gastelum CM, Plascencia-Aguilera LP, Arana-Nuno JR, Badillo-Camacho N, Marquez-Sandoval F, Holway FE, Vizmanos-Lamotte B. Anthropometric and Body Composition Profile of Young Professional Soccer Players. J Strength Cond Res. 2020 Jul;34(7):1911-1923. doi: 10.1519/JSC.0000000000003416. PMID 32058363
- [Background] Carvajal W, Rios A, Echevarria I, Martinez M, Minoso J, Rodriguez D. Body type and performance of elite cuban baseball players. MEDICC Rev. 2009 Apr;11(2):15-20. doi: 10.37757/MR2009V11.N2.6. PMID 21483313
- [Background] Dengel DR, Keller KA, Stanforth PR, Oliver JM, Carbuhn A, Bosch TA. Body Composition and Bone Mineral Density of Division 1 Collegiate Track and Field Athletes, a Consortium of College Athlete Research (C-CAR) Study. J Clin Densitom. 2020 Apr-Jun;23(2):303-313. doi: 10.1016/j.jocd.2019.07.008. Epub 2019 Jul 12. PMID 31399322
- [Background] Mangine GT, Mangine GT, Eggerth A, Gough J, Stratton MT, Feito Y, VanDusseldorp TA. Endocrine and Body Composition Changes Across a Competitive Season in Collegiate Speed-Power Track and Field Athletes. J Strength Cond Res. 2021 Aug 1;35(8):2067-2074. doi: 10.1519/JSC.0000000000004069. PMID 34100783
- [Background] Bonato M, Bizzozero S, Filipas L, LA Torre A. The influence of anthropometric parameters in track and field curve sprint. J Sports Med Phys Fitness. 2023 Dec;63(12):1254-1261. doi: 10.23736/S0022-4707.23.15056-0. Epub 2023 Aug 3. PMID 37535342
- [Background] Withers RT, Craig NP, Ball CT, Norton KI, Whittingham NO. The Drinkwater-Ross anthropometric fractionation of body mass: comparison with measured body mass and densitometrically estimated fat and fat-free masses. J Sports Sci. 1991 Autumn;9(3):299-311. doi: 10.1080/02640419108729891. PMID 1960800